CLINICAL TRIAL: NCT03701477
Title: Evaluation of the Efficacy of Trans-diagnostic Cognitive-behavioral Therapy on Controlling and Reducing Headache and Associated Symptoms Among Migrainous Patients
Brief Title: Trans-diagnostic Cognitive-behavioral Therapy for Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vahid Shaygannejad, Professor of Neurology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18820701962055
Record Dates: First submitted 2018-10-02; First posted 2018-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Migraine
Keywords: Migraine; trans-diagnostic approach; headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: control and intervention arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and outcomes assessors will be masked. The care provider and participants won't be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-diagnostic approach (Experimental): Trans-diagnostic cognitive-behavioral therapy In this arm, patients will participate in 10 sessions of therapy. During each session, specific topics will be discussed and participants will need to complete their homework for the next session. Each session lasts for 120 minutes. Sessions will be held in groups of 5-10 subjects weekly, except the last session that will be held after a two-week interval.
  Interventions: Behavioral: Trans-diagnostic cognitive-behavioral therapy
- Control (Sham Comparator): General relaxation/stress management therapeutic session In this arm, patients will attend a 3-hour meeting in which basic techniques of relaxation and overcoming stress and anxiety will be discussed.
  Interventions: Behavioral: General relaxation/stress management therapeutic session

INTERVENTIONS:
Behavioral: Trans-diagnostic cognitive-behavioral therapy — 10 therapeutic sessions hold in groups of 5-10 individuals. Details about each session: Session 1: Establishing rapport, psychoeducation; Session 2: Relaxation, hierarchy development; Session 3: Identifying automatic negative thoughts, guided imaginary; Session 4: Cognitive restructuring; Session 5: Problem solving skills training, distraction; Session 6: Exposure-based procedures, cognitive restructuring; Session 7-9: Advanced cognitive restructuring, stress management, assertiveness skills training, preparation for termination phase; Session 10: Relapse prevention, termination
  Arms: Trans-diagnostic approach
Behavioral: General relaxation/stress management therapeutic session — Patients will attend a 3-hour meeting in which basic techniques of relaxation and stress management will be discussed.
  Arms: Control

SUMMARY:
Migraine headache is one of the disabling conditions that may be associated with decreased quality of life, anxiety and depression. Currently, therapeutic approach to migraine is mostly based on prophylactic and acute phase medication therapy. Some investigators consider migraine a biopsychosocial condition which means that psychological therapies, such as cognitive-behavioral therapy and relaxation, may be efficient in controlling the disease. According to previous studies, cognitive therapies, including cognitive-behavioral therapy, have been efficient in decreasing frequency and severity of migraine, however, there are some challenges in applying these kind of interventions: the expenses; presence of multiple commodities that may lead to confusion and bewilderment for both therapist and patient; small number of trained psychologists for this intervention.

The trans-diagnostic approach, however, can facilitate some challenges with the previous method. Since it is not focused on a single condition, trained psychologists with this approach can apply it for a wide range of conditions, including migraine. Also, the trans-diagnostic approach leads to lower chances of confusion and bewilderment for therapist and patients. The trans-diagnostic approach focuses on therapeutic modules instead of constant similar therapeutic models. The five cores of trans-diagnostic approach are emotional awareness, cognitive flexibility, recognizing and preventing emotion avoidance and maladaptive emotion driven behaviors, awareness and tolerance of emotion-related physical conditions, and introceptive and situation-based emotion-focused exposure. This method was first designed to replace cognitive-behavioral therapy for emotional disorders, due to its feasibility and applicability.

The trans-diagnostic approach has been investigated by several researchers so far, however, most of those researches evaluate the efficacy of the technique on psychiatric disorders. It has also been investigated for treatment of headaches in adolescents. But no other study on other clinical problems or migraine has been conducted. Considering the high rates of comorbid anxiety and depressive symptoms in migrainous patients and the feasibility and efficacy of trans-diagnostic cognitive-behavioral therapy in other conditions, we aimed to evaluate its efficacy on controlling headache and related symptoms among migrainous patients.

DETAILED DESCRIPTION:
Migraine headache is one of the disabling conditions that occurs more in young women. It is usually associated with decreased quality of life, as well as anxiety and depressed in the affected individuals. Currently, therapeutic approach to migraine is mostly based on medication therapy in two phases of prophylaxis and acute attacks. However, some investigators consider it not only as a biologic disease, but also a multidimensional condition that may be accompanied by anxiety and depressive symptoms. Considering migraine as a biopsychosocial condition means that psychological therapies, such as cognitive-behavioral therapy and relaxation, may be efficient in controlling the disease. According to previous studies, cognitive therapies, including cognitive-behavioral therapy, have been efficient in decreasing frequency and severity of migraine, however, there are some challenges in applying these kind of interventions for patients: the costs of such treatments are usually not covered by insurance companies; presence of multiple commodities may lead to confusion and bewilderment for both therapist and patient while applying the technique; training psychologists for this intervention is costly and not enough psychologists know how to handle the condition.

The trans-diagnostic approach, however, can facilitate some challenges with the previous method. Since it is not focused on a single condition, trained psychologists with this approach can apply it for a wide range of conditions, including migraine. Also, the trans-diagnostic approach leads to lower chances of confusion and bewilderment for therapist and patients.

The trans-diagnostic approach is somehow similar to the classic cognitive-behavioral therapy. however, it focuses on therapeutic modules instead of constant similar therapeutic models. The five cores of trans-diagnostic approach are emotional awareness, cognitive flexibility, recognizing and preventing emotion avoidance and maladaptive emotion driven behaviors, awareness and tolerance of emotion-related physical conditions, and introceptive and situation-based emotion-focused exposure. This method was first designed to replace cognitive-behavioral therapy for emotional disorders, due to its feasibility and applicability.

The trans-diagnostic approach has been investigated by several researchers so far, however, most of those researches evaluate the efficacy of the technique on psychiatric disorders. It has also been investigated for treatment of headaches in adolescents. But no other study on other clinical problems or migraine has been conducted. Considering the high rates of comorbid anxiety and depressive symptoms in migrainous patients and the feasibility and efficacy of trans-diagnostic cognitive-behavioral therapy in other conditions, we aimed to evaluate its efficacy on controlling headache and related symptoms among migrainous patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine headache by primary neurologist based on the criteria defined by International Classification of Headache Disorders III Beta (ICHD-III Beta).
* Diagnosed with migraine at least 6 months prior to enrollment
* High school graduate or higher level of education

Exclusion Criteria:

* Medication overuse based on the criteria defined by ICHD-III Beta (taking non-steroidal anti-inflammatory drugs or other pain relievers at least 15 days in each month; taking triptans or similar drugs at least 10 days each month for 3 months or more)
* Addition of no new prophylactic migraine medication during the study
* suffering from other types of headache disorders
* Being treated with other psychological therapies (psychotherapy, ...) during the study.
* Not being able to fill our self-administered questionnaires (illiteracy, cognitive problems)
* Altered cognitive or mental status, like dementia

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before intervention; one month after the intervention
  Visual analog scale is used to rate the severity of headaches in patients. Patients are supposed to rate their pain on a scale from 0 to 10, 10 means the worst pain and 0 means no pain. They also can see cartoon faces that illustrate the severity of pain along with the numbers. Basically, lower numbers from this scale indicate better outcome. The scale has no sub-scale or other interpretation and the scores rated by patients will be described as the results.
Headache Impact Test-6 (HIT-6) | Before intervention; one month after the intervention
  This standard questionnaire evaluates the impact of headache on patient's ability to function on the job, at school, at home, or in social situations. It contains 6 questions (5-point Likert scale), each question covering one aspect of headache impact. The choices for each question can be never, rarely, sometimes, often, and always. These choices are rated as 6, 8, 10, 11, and 13 points, respectively, and the sum of scores shows the total score. The total score ranges from 36 (lowest score, the favorable outcome) to 78 (worst outcome, debilitating headaches). Also, scores higher than 50 mean that headache had caused significant disability for the patient. This questionnaire has no subscale and total scores will be reported.
Migraine Disability Assessment Scale (MIDAS) | Before intervention; one month after the intervention
  This standard questionnaire collects the days of disability due to headache. This questionnaire includes 5 questions, each question asking for number of the days that has caused a certain disability. The answers for these questions will be summed up to find the total score of the questionnaire. Based on the total score, the patient will be categorized in one of these groups: score 0-5 means no/unremarkable disability; score 6-10 means mild disability; score 11-20 means moderate disability; score>21 mean severe disability. As it was described, higher scores show worst outcome and lower scores present favorable outcome.
Hospital Anxiety and Depression Scale (HADS) | Before intervention; one month after the intervention
  This questionnaire evaluates general status of patient with respect to anxiety and depressive symptoms. The questionnaire contains 14 questions, 7 evaluate depression and 7 evaluate anxiety. Therefore, it has two subscales. Questions are 4-point Liker scales. Each question is scored from 0 to 3 based on the patient's choice, which is defined for each question. At the end, scores in each subscale are summed up to reach the total score on that subscale. In both subscales, score 0-7 means normal status, 8-10 means borderline status, and 11-21 means abnormal status on that subscale. As it was described, higher scores show worst outcome. The total score of the questionnaire won't be reported separately.

SECONDARY OUTCOMES:
Visual Analog Scale | Before intervention; Immediately after the intervention
  Visual analog scale is used to rate the severity of headaches in patients. Patients are supposed to rate their pain on a scale from 0 to 10, 10 means the worst pain and 0 means no pain. They also can see cartoon faces that illustrate the severity of pain along with the numbers. Basically, lower numbers from this scale indicate better outcome. The scale has no sub-scale or other interpretation and the scores rated by patients will be described as the results.
Headache Impact Test-6 (HIT-6) | Before intervention; Immediately after the intervention
  This standard questionnaire evaluates the impact of headache on patient's ability to function on the job, at school, at home, or in social situations. It contains 6 questions (5-point Likert scale), each question covering one aspect of headache impact. The choices for each question can be never, rarely, sometimes, often, and always. These choices are rated as 6, 8, 10, 11, and 13 points, respectively, and the sum of scores shows the total score. The total score ranges from 36 (lowest score, the favorable outcome) to 78 (worst outcome, debilitating headaches). Also, scores higher than 50 mean that headache had caused significant disability for the patient. This questionnaire has no subscale and total scores will be reported.
Migraine Disability Assessment Scale (MIDAS) | Before intervention; Immediately after the intervention
  This standard questionnaire collects the days of disability due to headache. This questionnaire includes 5 questions, each question asking for number of the days that has caused a certain disability. The answers for these questions will be summed up to find the total score of the questionnaire. Based on the total score, the patient will be categorized in one of these groups: score 0-5 means no/unremarkable disability; score 6-10 means mild disability; score 11-20 means moderate disability; score>21 mean severe disability. As it was described, higher scores show worst outcome and lower scores present favorable outcome.
Hospital Anxiety and Depression Scale (HADS) | Before intervention; Immediately after the intervention
  This questionnaire evaluates general status of patient with respect to anxiety and depressive symptoms. The questionnaire contains 14 questions, 7 evaluate depression and 7 evaluate anxiety. Therefore, it has two subscales. Questions are 4-point Liker scales. Each question is scored from 0 to 3 based on the patient's choice, which is defined for each question. At the end, scores in each subscale are summed up to reach the total score on that subscale. In both subscales, score 0-7 means normal status, 8-10 means borderline status, and 11-21 means abnormal status on that subscale. As it was described, higher scores show worst outcome. The total score of the questionnaire won't be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Shaygannejad, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Shokooh counselling center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
anonymized data will be made available upon request from researchers.

REFERENCES:
- [Result] Allen LB, Tsao JCI, Seidman LC, Ehrenreich-May J, Zeltzer LK. A Unified, Transdiagnostic Treatment for Adolescents With Chronic Pain and Comorbid Anxiety and Depression. Cogn Behav Pract. 2012 Feb;19(1):56-67. doi: 10.1016/j.cbpra.2011.04.007. PMID 28824271
- [Result] Bullis JR, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Carl JR, Barlow DH. The unified protocol for transdiagnostic treatment of emotional disorders: preliminary exploration of effectiveness for group delivery. Behav Modif. 2015 Mar;39(2):295-321. doi: 10.1177/0145445514553094. Epub 2014 Oct 14. PMID 25316034
- [Result] Buse DC, Rupnow MF, Lipton RB. Assessing and managing all aspects of migraine: migraine attacks, migraine-related functional impairment, common comorbidities, and quality of life. Mayo Clin Proc. 2009 May;84(5):422-35. doi: 10.1016/S0025-6196(11)60561-2. PMID 19411439
- [Result] D'Amico D, Leonardi M, Grazzi L, Curone M, Raggi A. Disability and quality of life in patients with different forms of migraine. J Headache Pain. 2015 Dec;16(Suppl 1):A4. doi: 10.1186/1129-2377-16-S1-A4. No abstract available. PMID 28132384
- [Result] Harris P, Loveman E, Clegg A, Easton S, Berry N. Systematic review of cognitive behavioural therapy for the management of headaches and migraines in adults. Br J Pain. 2015 Nov;9(4):213-24. doi: 10.1177/2049463715578291. PMID 26526604
- [Result] Myhr G, Payne K. Cost-effectiveness of cognitive-behavioural therapy for mental disorders: implications for public health care funding policy in Canada. Can J Psychiatry. 2006 Sep;51(10):662-70. doi: 10.1177/070674370605101006. PMID 17052034
- [Result] Norton PJ, Barrera TL. Transdiagnostic versus diagnosis-specific cbt for anxiety disorders: a preliminary randomized controlled noninferiority trial. Depress Anxiety. 2012 Oct;29(10):874-82. doi: 10.1002/da.21974. Epub 2012 Jul 5. PMID 22767410
- [Result] Singer AB, Buse DC, Seng EK. Behavioral treatments for migraine management: useful at each step of migraine care. Curr Neurol Neurosci Rep. 2015 Apr;15(4):14. doi: 10.1007/s11910-015-0533-5. PMID 25708673
- [Result] Sullivan A, Cousins S, Ridsdale L. Psychological interventions for migraine: a systematic review. J Neurol. 2016 Dec;263(12):2369-2377. doi: 10.1007/s00415-016-8126-z. Epub 2016 May 9. PMID 27159991
- [Derived] Soleimanian-Boroujeni F, Badihian N, Badihian S, Shaygannejad V, Gorji Y. The efficacy of transdiagnostic cognitive behavioral therapy on migraine headache: a pilot, feasibility study. BMC Neurol. 2022 Jun 22;22(1):230. doi: 10.1186/s12883-022-02729-8. PMID 35733127